CLINICAL TRIAL: NCT00732693
Title: Comparison of Standard and Physiologic Sex Steroid Replacement Regimens in Women With Premature Ovarian Failure and the Assessment of Skeletal, Cardiovascular and Reproductive Parameters
Brief Title: Evaluation of Physiologic and Standard Sex Steroid Replacement Regimens in Women With Premature Ovarian Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Edinburgh (Other)
Responsible Party: Dr W Hamish B Wallace, Consultant/Reader in Paediatric Oncology, NHS Lothian / University of Edinburgh
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CLIC/Sargent-178000-R35464
Record Dates: First submitted 2008-08-11; First posted 2008-08-12 (Estimated); Last update posted 2008-08-12 (Estimated); Status verified 2008-08

CONDITIONS: Premature Ovarian Failure
Keywords: Premature ovarian failure; Sex hormone replacement; HRT; Blood pressure; Bone mineral density; Bone metabolism; Uterine function
MeSH Terms: conditions — Primary Ovarian Insufficiency | interventions — Ethinyl Estradiol; Norethindrone; Estradiol; Progesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Treatment with standard sex steroid replacement regimen
  Interventions: Drug: Ethinylestradiol / Norethisterone
- 2 (Experimental): Treatment with physiologic sex steroid regimen
  Interventions: Drug: Estradiol / Progesterone

INTERVENTIONS:
Drug: Ethinylestradiol / Norethisterone — Oral ethinylestradiol 30mcg and norethisterone 1.5mg daily for weeks 1-3, followed by 7 "pill free" days
  Other Names: Loestrin 30, Galen Ltd, UK
  Arms: 1
Drug: Estradiol / Progesterone — Transdermal estradiol 100mcg daily for week 1, then 150mcg daily for weeks 2-4; and vaginal progesterone pessaries 200mg twice daily for weeks 3-4
  Other Names: Estraderm TTS, Novartis Pharmaceuticals UK Ltd; Cyclogest, Activis UK Ltd
  Arms: 2

SUMMARY:
The aim of the study is to determine whether physiological sex steroid replacement improves parameters of skeletal, cardiovascular and reproductive health of women treated with current sex steroid replacement regimens.

DETAILED DESCRIPTION:
Premature ovarian failure, defined as the onset of the menopause before the age of 40 years, is a relatively common problem that affects 1% of women. There are a variety of aetiologies underlying premature ovarian failure including Turner syndrome and those with idiopathic onset, however with the increasing success of intensive treatment for childhood cancer, there are increasing numbers of young survivors, with a variety of late effects of treatment, including premature ovarian failure.

Evidence is required for the optimal management of young women with premature ovarian failure, either as a result of childhood cancer treatment or for other reasons. These women are currently offered combined sex steroid replacement in the convenient form of the oral contraceptive pill, or hormone replacement therapy, designed for older women after the menopause. These preparations are not designed to achieve physiological replacement of oestrogen or progesterone, either in dosage or in biochemical structure - many preparations using synthetic derivatives. These younger women who have differing metabolic and psychological requirements are looking to a future of 30 or more years of replacement. The optimal mode of SSR is not known for young women with premature ovarian failure, however there is concern that current regimens may be inadequate for optimal skeletal and cardiovascular health.

Current preliminary data demonstrates that use of physiological sex steroid replacement improves uterine parameters. Evidence is required to determine whether optimising sex steroid replacement can also significantly improve parameters of skeletal and cardiovascular health. Young women with ovarian failure face several decades of hormone replacement, so small improvements in management may make large differences to later morbidity and mortality.

The aim of the study is to determine whether physiological sex steroid replacement improves parameters of skeletal, cardiovascular and reproductive health of women treated with current sex steroid replacement regimens.

ELIGIBILITY:
Inclusion Criteria:

* Premature Ovarian Failure

Exclusion Criteria:

* Intercurrent illness

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2002-02; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Change in 24 hour ambulatory blood pressure | Before each washout period, then at 0, 3, 6 and 12 months of each treatment
Bone mineral density measurements (DEXA) | Baseline, 14 and 24 months
Uterine ultrasound scan to assess uterine volume, endometrial thickness, and uterine artery blood flow | Before each washout period, then at 0, 3, 6 and 12 months of each treatment

SECONDARY OUTCOMES:
Central arterial blood pressure and arterial stiffness measured using peripheral arterial tonometry | Before each washout period, then at 0, 3, 6 and 12 months of each treatment phase
Biochemical evidence of activity on the renin-angiotensin system, including plasma renin activity, angiotensin II, aldosterone, creatinine, urea and electrolyte concentrations. | Before each washout period, then at 0, 3, 6 and 12 months of each treatment phase
Serum markers of collagen turnover and bone matrix formation | Before each washout period, then at 0, 3, 6 and 12 months of each treatment phase
Hormonal assays for gonadotrophins, FSH, LH and sex steroids estrogen and progesterone | Before each washout period, then at 0, 3, 6 and 12 months of each treatment phase

CONTACTS AND LOCATIONS:
Overall Officials: W Hamish B Wallace, MD, Principal Investigator — NHS Lothian / University of Edinburgh
Locations (2):
- United Kingdom (2):
  - Royal Infirmary of Edinburgh, Edinburgh
  - Royal Hospital for Sick Children, Edinburgh

REFERENCES:
- [Background] Bath LE, Critchley HO, Chambers SE, Anderson RA, Kelnar CJ, Wallace WH. Ovarian and uterine characteristics after total body irradiation in childhood and adolescence: response to sex steroid replacement. Br J Obstet Gynaecol. 1999 Dec;106(12):1265-72. doi: 10.1111/j.1471-0528.1999.tb08180.x. PMID 10609720
- [Background] Critchley HO, Buckley CH, Anderson DC. Experience with a 'physiological' steroid replacement regimen for the establishment of a receptive endometrium in women with premature ovarian failure. Br J Obstet Gynaecol. 1990 Sep;97(9):804-10. doi: 10.1111/j.1471-0528.1990.tb02574.x. PMID 2242365
- [Background] Critchley HO, Wallace WH, Shalet SM, Mamtora H, Higginson J, Anderson DC. Abdominal irradiation in childhood; the potential for pregnancy. Br J Obstet Gynaecol. 1992 May;99(5):392-4. doi: 10.1111/j.1471-0528.1992.tb13755.x. PMID 1622911
- [Background] Davies MC, Gulekli B, Jacobs HS. Osteoporosis in Turner's syndrome and other forms of primary amenorrhoea. Clin Endocrinol (Oxf). 1995 Dec;43(6):741-6. doi: 10.1111/j.1365-2265.1995.tb00544.x. PMID 8736278
- [Background] Hansen SW, Olsen N. Raynaud's phenomenon in patients treated with cisplatin, vinblastine, and bleomycin for germ cell cancer: measurement of vasoconstrictor response to cold. J Clin Oncol. 1989 Jul;7(7):940-2. doi: 10.1200/JCO.1989.7.7.940. PMID 2472472
- [Background] Hawkins MM, Smith RA. Pregnancy outcomes in childhood cancer survivors: probable effects of abdominal irradiation. Int J Cancer. 1989 Mar 15;43(3):399-402. doi: 10.1002/ijc.2910430309. PMID 2538400
- [Background] Hoorweg-Nijman JJ, Kardos G, Roos JC, van Dijk HJ, Netelenbos C, Popp-Snijders C, de Ridder CM, Delemarre-van de Waal HA. Bone mineral density and markers of bone turnover in young adult survivors of childhood lymphoblastic leukaemia. Clin Endocrinol (Oxf). 1999 Feb;50(2):237-44. doi: 10.1046/j.1365-2265.1999.00654.x. PMID 10396368
- [Background] Howell SJ, Shalet SM. Aetiology-specific effect of premature ovarian failure on bone mass - is residual ovarian function important? Clin Endocrinol (Oxf). 1999 Nov;51(5):531-4. doi: 10.1046/j.1365-2265.1999.00891.x. No abstract available. PMID 10594512
- [Background] Kaneko N, Kawagoe S, Hiroi M. Turner's syndrome--review of the literature with reference to a successful pregnancy outcome. Gynecol Obstet Invest. 1990;29(2):81-7. doi: 10.1159/000293307. PMID 2185981
- [Background] Krolner B, Pors Nielsen S. Bone mineral content of the lumbar spine in normal and osteoporotic women: cross-sectional and longitudinal studies. Clin Sci (Lond). 1982 Mar;62(3):329-36. doi: 10.1042/cs0620329. PMID 6977427
- [Background] Mendelsohn ME, Karas RH. The protective effects of estrogen on the cardiovascular system. N Engl J Med. 1999 Jun 10;340(23):1801-11. doi: 10.1056/NEJM199906103402306. No abstract available. PMID 10362825
- [Background] Register TC, Jayo MJ, Jerome CP. Oral contraceptive treatment inhibits the normal acquisition of bone mineral in skeletally immature young adult female monkeys. Osteoporos Int. 1997;7(4):348-53. doi: 10.1007/BF01623776. PMID 9373569
- [Background] Rubin K. Turner syndrome and osteoporosis: mechanisms and prognosis. Pediatrics. 1998 Aug;102(2 Pt 3):481-5. PMID 9685448
- [Background] Saenger P. Clinical review 48: The current status of diagnosis and therapeutic intervention in Turner's syndrome. J Clin Endocrinol Metab. 1993 Aug;77(2):297-301. doi: 10.1210/jcem.77.2.8345029. No abstract available.
- [Derived] O'Donnell RL, Warner P, Lee RJ, Walker J, Bath LE, Kelnar CJ, Wallace WH, Critchley HO. Physiological sex steroid replacement in premature ovarian failure: randomized crossover trial of effect on uterine volume, endometrial thickness and blood flow, compared with a standard regimen. Hum Reprod. 2012 Apr;27(4):1130-8. doi: 10.1093/humrep/des004. Epub 2012 Feb 16. PMID 22343553